CLINICAL TRIAL: NCT04335786
Title: PRAETORIAN-COVID: A Double-blind, Placebo-controlled Randomized Clinical Trial With Valsartan for PRevention of Acute rEspiraTORy dIstress Syndrome in hospitAlized patieNts With SARS-COV-2 (COVID-19) Infection Disease
Brief Title: Valsartan for Prevention of Acute Respiratory Distress Syndrome in Hospitalized Patients With SARS-COV-2 (COVID-19) Infection Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment was stopped to facilitate successful enrollment for the ACE2RAS-domain of the REMAP-CAP trial.
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL73547.091.20; 2020-001320-34 (EudraCT Number)
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2020-04

CONDITIONS: Acute Respiratory Distress Syndrome; SARS-CoV-2; COVID; COVID-19; Severe Acute Respiratory Syndrome
Keywords: Acute Respiratory Distress Syndrome; SARS-CoV-2; Therapeutics; Valsartan; Angiotensin Receptor Blockade; Angiotensin Receptor Blockers; ARBs; COVID-19
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19; Severe Acute Respiratory Syndrome | interventions — Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active treatment arm (Experimental): Valsartan at a dosage and frequency titrated to blood pressure with 80mg or 160mg tablets up to a maximum dose of 160mg b.i.d.
  Interventions: Drug: Valsartan (Diovan)
- Placebo arm (Placebo Comparator): Matching 80mg or 160mg placebo tablets at a dosage and frequency titrated to systolic blood pressure
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Valsartan (Diovan) — At the time of randomization each participant will start with study treatment and continue up to 14 days, or up to reaching the primary endpoint, or up to hospital discharge, or up to any of the pre-defined stopping criteria.
  Study drug dosages will be titrated to blood pressure with a maximum of 160mg b.i.d.
  Arms: Active treatment arm
Drug: Placebo oral tablet — At the time of randomization each participant will start with study treatment and continue up to 14 days, or up to reaching the primary endpoint, or up to hospital discharge, or up to any of the pre-defined stopping criteria.
  Arms: Placebo arm

SUMMARY:
Rationale: The current SARS-CoV-2 pandemic has a high burden of morbidity and mortality due to development of the so-called acute respiratory distress syndrome (ARDS). The renin-angiotensin-system (RAS) plays an important role in the development of ARDS.

ACE2 is one of the enzymes involved in the RAS cascade. Virus spike protein binds to ACE2 to form a complex suitable for cellular internalization. The downregulation of ACE2 results in the excessive accumulation of angiotensin II, and it has been demonstrated that the stimulation of the angiotensin II type 1a receptor (AT1R) increases pulmonary vascular permeability, explaining the increased lung pathology when activity of ACE2 is decreased. Currently available AT1R blockers (ARBs) such as valsartan, have the potential to block this pathological process mediated by angiotensin II. There are presently two complementary mechanisms suggested: 1) ARBs block the excessive angiotensin-mediated AT1R activation, and 2) they upregulate ACE2, which reduces angiotensin II concentrations and increases the production of the protective vasodilator angiotensin 1-7. In light of the above, ARBs may prevent the development of ARDS and avert morbidity (admission to intensive care unit (ICU) and mechanical ventilation) and mortality.

Objective: To investigate the effect of the ARB valsartan in comparison to placebo on the occurrence of one of the following items, within 14 days of randomization:1) ICU admission; 2) Mechanical ventilation; 3) Death.

Study design: A double-blind, placebo-controlled 1:1 randomized clinical trial Study population: Adult hospitalized SARS-CoV-2-infected patients (n=651). Intervention: The active-treatment arm will receive valsartan in a dosage titrated to blood pressure up to a maximum of 160mg b.i.d. and the placebo arm will receive a matching placebo also titrated to blood pressure. Treatment duration will be 14 days or up to hospital discharge < 14 days or occurrence of the primary endpoint if < 14 days.

Main study endpoint: The primary study endpoint is the occurrence within 14 days of randomization of either: 1) ICU admission; 2) Mechanical ventilation; 3) Death.

ELIGIBILITY:
Inclusion Criteria

* Adult (age ≥ 18 years)
* Admitted to the hospital of any participating center
* Confirmed SARS-CoV-2 infection with either: positive laboratory test for SARS-CoV-2* ; or positive CT thorax diagnostic for SARS-CoV-2 infection according to the prevailing criteria
* Randomization:

  * Within 24 hours of confirmed in-hospital SARS-CoV-2 infection diagnosis OR
  * within 24 hours of hospital admission in case of pre-hospital confirmed SARS-CoV-2 infection.

    * In case there is a lack of laboratory tests for SARS-CoV-2 in the participating center of the potentially eligible patient, a positive laboratory test for SARS-CoV-2 will be no longer required. In that case, the potentially eligible patient needs to meet the prevailing criteria for the diagnosis of SARS-CoV-2 infection of that participating center, such as typical abnormalities on pulmonary CT in the setting of high clinical suspicion of SARS-CoV-2 infection.

Exclusion Criteria:

* Admitted to ICU prior to randomization
* Currently taking an ARB or angiotensin-receptor-neprilysin-inhibitor (ARNI)
* Use of other investigational drugs at the time of enrollment
* Prior reaction or intolerance to an ARB or ARNI; or severe intolerance to an ACEi, defined as angio-oedema requiring medical intervention
* Systolic blood pressure < 105mmHg or diastolic blood pressure <65mmHg
* Potassium greater than 5.5 mEq/L within 4 weeks of study enrollment.
* Estimated Glomerular Filtration Rate (eGFR) of < 30ml/min/1.73 m2 within 4 weeks of study initiation
* A known history of renal artery stenosis
* AST and/or ALT > 3 times the upper limit of normal within 4 weeks of study enrollment. In case of mild to moderate liver dysfunction valsartan dosage will be limited to a maximum of 80mg
* Severe liver dysfunction, biliary cirrhosis or cholestasis
* Severe volume depletion or severe acute kidney injury that, in the opinion of the investigator, would preclude administration of valsartan
* Concurrent treatment with Aliskiren
* Inability to obtain informed consent
* Pregnancy or breastfeeding
* In females of childbearing age, unwillingness to use birth control or to be sexually abstinent for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
first occurrence of intensive care unit admission, mechanical ventilation or death | within 14 days
  Death is defined as all-cause mortality

SECONDARY OUTCOMES:
Death | Within 14 days, 30 days, 90 days and at 1 year
  All-cause mortality; and time to all-cause mortality
Mechanical ventilation | within 14 days
  Occurrence of mechanical ventilation and time to ventilation
Intensive care unit admission | within 14 days
  Occurrence of ICU admission and time to admission
Occurrence of acute kidney injury | Within 14 days
  Defined as a 50% decline in estimated glomerular filtration rate relative to baseline, or decrease of >30 ml/min/1.73m2 and to a value below 60 ml/min/1.73m2

CONTACTS AND LOCATIONS:
Overall Officials: Niels van Royen, MD PhD, Study Chair — Radboud University Medical Center
Locations (7):
- Netherlands (7):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Rijnstate, Arnhem
  - Radboudumc, Nijmegen
  - Laurentius Ziekenhuis, Roermond
  - Erasmus MC, Rotterdam
  - Franciscus Gasthuis, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam

REFERENCES:
- [Derived] Gommans DHF, Nas J, Pinto-Sietsma SJ, Koop Y, Konst RE, Mensink F, Aarts GWA, Konijnenberg LSF, Cortenbach K, Verhaert DVM, Thannhauser J, Mol JQ, Rooijakkers MJP, Vos JL, van Rumund A, Vart P, Hassing RJ, Cornel JH, de Jager CPC, van den Heuvel MM, van der Hoeven HG, Verbon A, Pinto YM, van Royen N, van Kimmenade RRJ; Event committee; de Leeuw PW, van Agtmael MA, Bresser P; Data Safety Monitoring Board; van Gilst WH, Vonk-Noordergraaf A, Tijssen JGP; Steering committee; van Royen N, de Jager CPC, van den Heuvel MM, van der Hoeven HG, Verbon A, Pinto YM, van Kimmenade RRJ. Rationale and design of the PRAETORIAN-COVID trial: A double-blind, placebo-controlled randomized clinical trial with valsartan for PRevention of Acute rEspiraTORy dIstress syndrome in hospitAlized patieNts with SARS-COV-2 Infection Disease. Am Heart J. 2020 Aug;226:60-68. doi: 10.1016/j.ahj.2020.05.010. Epub 2020 May 21. PMID 32512291